CLINICAL TRIAL: NCT05950373
Title: Educational Intervention for Better Nutrition to Preserve Functionality - Design of a Randomised Clinical Trial
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Nord University (Other)
Responsible Party: Principal Investigator, Monica Christin Hansen, PhD student, Nord University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 366925
Record Dates: First submitted 2023-07-11; First posted 2023-07-18 (Actual); Last update posted 2024-04-03 (Actual); Status verified 2024-04

CONDITIONS: Malnutrition
Keywords: Older adults; Diseases-related malnutrition; Educational video
MeSH Terms: conditions — Malnutrition

STUDY DESIGN:
Who Masked: Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental): The Intervention group will get access to a six-minute long education video five days after being discharges from the hospital. The video is focusing on protein and energy meals for older adults.
  The educational film is available via a link on a tablet/ computer or mobile phone.
  The education video vil only be given one time.
  Interventions: Other: Education video
- Control group (No Intervention): The control group will not be given any intervention.

INTERVENTIONS:
Other: Education video — six minute long education video focusing on protein and energy meals for older adults.
  Arms: Intervention group

SUMMARY:
This project explores whether access to a digital education video can improve the nutritional situation of home-living older adults after being discharged from the hospital.

ELIGIBILITY:
Inclusion Criteria:

* Surgical patients embedded in a regional hospital.
* Home-living in one of nine selected municipalities.
* Be able to read and understand Norwegian.
* Have a consent competence.
* Have a body mass index < 24.
* Have access to a digital solution such as a tablet or phone.

Exclusion Criteria:

* Persons given only a liquid diet.
* Persons in a terminally ill phase.

Ages: 65 Years to 110 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 276 (Estimated)
Dates: Start 2025-01-01 (Estimated); Primary Completion 2025-11-30 (Estimated); Study Completion 2026-10-01 (Estimated)

PRIMARY OUTCOMES:
Health related quality of life Using Rand 36 questionaire | Change in Health related quality of life Using Rand 36 questionaire after 3 months
  Using Rand 36 questionaire. The data from the SF-36 ordinal subscales will be transformed to a ratio scale using the syntax SF-36 manual and will be presented as the results from each of the eight subscales and the two main scales

SECONDARY OUTCOMES:
Body fat | Change in Body mass index after 3 months.
  Body fat will be measured by Body mass index (BMI). Weight (in kg) and height (in cm) will be combined to report BMI in Kg/m2
Readmissions to hospital after discharge from the hospital | Registration of Readmissions 3 months after
  Readmissions after discharge from the hospital will be measured three months after discharge.
Muscle strength | Change in Hand Grip Strength (muscle strength) after 3 months
  Measure Muscle Strength (in Kg) using Hydraulic Hand dynameter for Hand Grip strength in both hands.
The mid-arm circumferences | Change in the mid-arm cirumferences after three months.
  The mid-arm circumferences (MAC) will be measured in cm with a measuring tape. This will be done on the left upper arm measured at the midpoint between the top of the shoulder and the tip of the elbow.
Subcutaneous fat | Change in Subcutaneous fat after three months.
  Subcutaneous fat will be measured by Triceps skinfold thickness (TFS). This will be done in millimetres with a VirtuFits Digital Fat caliper skinfold in the triceps of the left arm.
Muscle protein mass | Change in Muscle protein mass after 3 months
  Muscle protein mass will be measured by the mean arm muscle circumferences (MAMC) calculated to the formula: MAMC (cm) = MAC (cm) - (3,14 X TFS X 0,1)
Knowledge about nutrition | Registration in a questionaire three months after discharge from the hospital.
  Participants' knowledge about nutrition will be measured with a questionaire consisting of three questions related to the education video.

CONTACTS AND LOCATIONS:
Locations (1):
- Monica Christin Hansen, Bodø, Norway

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Hansen MC, Uhrenfeldt L, Ingstad K, Pedersen PU. Educational nutritional intervention to prevent loss of health-related quality of life among older adults after a surgical treatment: design of a randomised controlled trial. Trials. 2024 Apr 15;25(1):262. doi: 10.1186/s13063-024-08096-8. PMID 38622729